CLINICAL TRIAL: NCT03178630
Title: Longitudinal Study for the Assessment of MRI Based Biomarkers as a Predictors of Clinical Endpoints in Pediatric Onset Autoimmune Liver Disease
Brief Title: MRI Biomarkers in as Predictor of Clinical Endpoints in Pediatric Autoimmune Liver Disease
Status: Recruiting | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: CIN002 MRI biomarkers in AILD
Record Dates: First submitted 2017-03-30; First posted 2017-06-07 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Liver Disease; Autoimmune Hepatitis; Primary Sclerosing Cholangitis
MeSH Terms: conditions — Hepatitis, Autoimmune; Cholangitis, Sclerosing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma and serum samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with autoimmune liver disease: Patients with autoimmune liver disease
  Patients (6-23 y.o.) with established clinical diagnosis of AIH or suspected diagnosis of AIH based on elevated serum AST or ALT, elevated IgG level >1.1 ULN, elevated titer of autoantibodies, including ANA, SMA, LKM, LC-1 or SLA, which is consistent with the simplified criteria for the diagnosis of AIH in children will be enrolled.
  Patients (6-23 y.o.) with established clinical diagnosis of PSC or Suspected diagnosis of PSC supported by abnormal cholangiogram (ERCP or MRCP) or elevated GGT>1.5 ULN and dilated bile ducts by liver ultrasound will be enrolled.

SUMMARY:
Autoimmune liver diseases (AILD), which include Primary Sclerosing Cholangitis (PSC) and Autoimmune Hepatitis (AIH) are a common etiological factor for chronic liver disease among adolescents. This is a longitudinal study to identify surrogate endpoints with an accurate predictive value for the progression of hepatobiliary damage in subjects with pediatric onset AILD. This study will involve collection of MRI-based data at the time of enrollment and at year 1 and 2 of follow up, and collection of clinical data for 10 years following enrollment. There is a strong possibility that MRI quantitative techniques may be more sensitive to disease progression than standard clinical and laboratory tests. To investigate predictivity of MRI based biomarkers, summary measures of MRCP/MREL from baseline, Year 1 and Year 2, e.g. change rate, maximum, and average will be calculated as predictors for Year 10 clinical outcomes. The same predictors will also be used to model native liver survival in a proportional hazard regression. Findings from this study may be used to assess disease progression and to predict complications and survival of liver disease patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age 6-23 years old.
2. Established clinical diagnosis of AIH or PSC.

Exclusion Criteria:

1. History of liver transplantation.
2. Chronic Hepatitis B or untreated hepatitis C virus infection.
3. Pregnancy.
4. Absolute contraindication for MRI (e.g. pacemaker, metallic implants, claustrophobia).
5. Diagnosis of cystic fibrosis or biliary atresia
6. Diagnosis of cardiac hepatopathy.
7. Diagnosis of Wilson's disease, Alpha-1 Antitrypsin deficiency, or Glycogen storage disease.
8. Skin conditions which could be aggravated by MREL (i.e. Epidermolysis bullosa).

Ages: 6 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 150 patients between 6 and 23 years of age with a diagnosis of PSC or AIH will be enrolled and followed up to 10 Years.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2017-02-20 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2031-02 (Estimated)

PRIMARY OUTCOMES:
Change of intrahepatic bile duct irregularities between V0 (baseline visit) and V1 (visit after12 months) or V2 (visit after 24 months). | 24 months
  Change of intrahepatic bile duct irregularities between V0 and V1 or V2 by MRCP (scored by Majoie classification on 4 point scale of 0-3).
Change of extra-hepatic duct irregularities between V0 (baseline visit) and V1 (visit after 12 months) or V2 (visit after 24 months). | 24 months
  Change of extra-hepatic duct irregularities between V0 and V1 or V2 by MRCP (scored by Majoie classification on 5 point scale 0-4).
Mean shear stiffness of the liver | 24 months
  Change in mean shear stiffness (kPa) of the liver by MREL between V0 (baseline visit) and V1 ( visit after 12 months) or V2 (visit after 24 months).
long-term clinical outcomes: survival with the native liver | 120 months
  Annual assessment of survival with the native liver (Yes=1, No=0) will be done within 10 years of follow-up.
long-term clinical outcomes: hospital admissions for cholangitis | 120 months
  Annual assessment of long-term clinical outcomes will be done within 10 years of follow-up. Any hospital admissions for cholangitis (Yes=1, No=0) since last visit will be recorded at the time of follow-up.
long-term clinical outcomes:endoscopic interventions for biliary strictures | 120 months
  Annual assessment of long-term clinical outcomes will be done within 10 years of follow-up. Endoscopic interventions for biliary strictures (Yes=1, No=0) since last visit will be recorded at the time of follow-up.
long-term clinical outcomes:diagnosis of cholangiocarcinoma | 120 months
  Annual assessment of long-term clinical outcomes will be done within 10 years of follow-up. If there is diagnosis of cholangiocarcinoma (Yes=1, No=0) since last visit will be recorded.
long-term clinical outcomes: variceal bleeding | 120 months
  Annual assessment of long-term clinical outcomes will be done within 10 years of follow-up. Presence or absence of variceal bleeding (Yes=1, No=0) since last visit will be recorded.
long-term clinical outcomes: ascites | 120 months
  Annual assessment of long-term clinical outcomes will be done within 10 years of follow-up. Presence or absence of ascites (Yes=1, No=0) since last visit will be recorded.

SECONDARY OUTCOMES:
Changes in liver/spleen volumes | 24 months
  Changes in liver/spleen volumes (mL) between V0 (baseline visit) and V1 (visit after 12 months) or V2 (visit after 24 months).
Changes in T1rho, T1 and T2 mapping | 24 months
  Readouts of T1rho, T1 and T2 mapping between baseline MRI at V0 (baseline visit) and repeat ones at V1 (after12 months) or V2 (after 24 months) in msec.
Clinical endpoints of AILD: Pruritus | 120 months
  Annual assessment for Pruritus (on visual analogue scale of 0-10) will be done within 10 years of follow-up.
Clinical endpoints of AILD | 120 months
  Annual assessment for Clinical diagnosis of hepatopulmonary syndrome (Yes=1, No=0) and/or hepatic encephalopathy (Yes=1, No=0) will be done within 10 years of follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Alexander Miethke, MD, Principal Investigator — Cincinnati Childrens Hospital Medical Center
Locations (1):
- Cincinnati Children's Hospital and Medical Center, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No